CLINICAL TRIAL: NCT00301249
Title: The Family Investigation of Nephropathy and Diabetes (FIND) Study
Brief Title: The Family Investigation of Nephropathy and Diabetes Study
Acronym: FIND
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Case Western Reserve University (Other)
Responsible Party: Sponsor
Other Study IDs: FIND U01DK057292; U01DK057292 (NIH)
Record Dates: First submitted 2006-03-09; First posted 2006-03-10 (Estimated); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Diabetes; Diabetic Nephropathy
Keywords: Diabetes; Nephropathy; Diabetic Nephropathy; Genome Scan; Genetic Research
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Nephropathies; Kidney Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Family Investigation of Nephropathy and Diabetes (FIND): Individuals with diabetic nephropathy, their parents, and selected siblings
- African American MALD: Case-control study of African American patients with nephropathy (cases) and their spouses (controls) unaffected by diabetes and nephropathy; offspring were genotyped when available to provide haplotype data.
- Mexican American MALD: Case-control study of unrelated individuals of Mexican American heritage in which both cases and controls had diabetes, but only the case had nephropathy

SUMMARY:
The Family Investigation of Nephropathy and Diabetes (FIND)Study is a multi-center consortium. The charge of the consortium is to acquire sets of families with well-characterized diabetic nephropathy, establish a secure master FIND database, and perform a genome scan to identify chromosomal regions linked with diabetic nephropathy.

DETAILED DESCRIPTION:
Diabetic Nephropathy (DN) is undoubtedly a multifactorial disease, and a large proportion of patients affected with either type 1 or type 2 diabetes develop diabetic nephropathy and progress to end stage renal disease (ESRD). When poor prognostic factors such as hypertension and chronic hyperglycemia are aggressively treated, the rate of progression of diabetic nephropathy can be slowed. However, no interventions have been shown to reliably halt the progression of diabetic nephropathy. Numerous studies have suggested that genetic predisposition to diabetic nephropathy exists, but genes for nephropathy have not yet been isolated. It is anticipated that a comprehensive analysis of a large number of uniformly phenotyped ESRD families will be necessary to isolate genes for ESRD. Such a database of families may not be available at any single institution. The FIND study has established a centralized Genetic Analysis and Data Coordinating Center (GADCC) that, together with eight participating investigation centers (PICs), three minority recruitment centers, and the National Institute of Diabetes, Digestive and Kidney Diseases (NIDDK), will use the emerging high-throughput genetic technologies to enable identification of diabetic nephropathy susceptibility or protection genes. The charge of the consortium is to acquire sets of families with well-characterized diabetic nephropathy, establish a secure master FIND database, and perform a genome scan to identify chromosomal regions linked with diabetic nephropathy. The FIND study population includes participants from European American (EA), Native American (NA), African American (AA) and Mexican American (AA) populations.

Two analytic approaches are utilized in FIND. The Family Study approach involves the enrollment of probands, affected or discordant sibling and their affected family members. Analytic methods include affected sibling pair (ASP), discordant sibling pair (DSP) affected relative pair (ARP), and discordant relative pair (DRP) linkage analyses for the Family Study. The Mapping by Admixture and Linkage Disequilibrium (MALD) approach involves the enrollment of probands and a population based control for both the AA and MA studies. In addition, a spousal control (diad) and when available, a child 18 years or older, will be recruited (triad)for the AA MALD study only.

ELIGIBILITY:
Inclusion Criteria:

For the Family protocol, proband must meet diagnostic criteria for diabetes and have nephropathy that meets one of the following:

* diabetic nephropathy diagnosed from a kidney biopsy and a history of overt proteinuria.
* ESRD considered due to diabetic nephropathy because
* diabetes is present for ≥ 5 years prior to the initiation of renal replacement therapy and diabetic retinopathy has been diagnosed at any time; or
* diabetes is present ≥ 5 years prior to the initiation of replacement therapy and either a 24 hour urine collection contains ≥ 3 gm protein/24 hours or a random urine protein (mg/dl)/ creatinine (mg/dl) ratio is ≥ 3.0; or
* diabetic retinopathy is present and either a previous 24 hour urine collection contains ≥ 3 gm protein/24 hours or a random urine protein (mg/dl)/ creatinine (mg/dl) ratio is ≥ 3.0.
* nephropathy without ESRD that is considered to be diabetic nephropathy because (a) diabetic retinopathy and a 24 hr urine collection with either ≥ 1 gram proteinuria/24 hours or a urine protein (mg/dl)/ creatinine (mg/dl) ratio ≥ 1.0; or (b) at a time when diabetes duration is ≥ 10 years, either a urine collection of ≥ 3 grams protein/24 hours or a urine protein (mg/dl) /creatinine (mg/dl) ratio ≥ 3.0.

African-American patients with chronic renal failure are as MALD cases by meeting criteria for diabetic nephropathy, as described for Family probands, or having nephropathy (serum creatinine ≥ 2.0 mg/dl) not due to diabetes or known monogenic renal disease. Mexican-Americans recruited as MALD cases must meet criteria for diabetic nephropathy as defined for the Family probands. Phenotype criteria for probands entered into the Family or MALD protocols must be confirmed by medical record review.

Eligibility of family members and MALD control subjects is based on laboratory tests obtained at the time of screening. Entry of a proband with diabetic nephropathy into the Family protocol also requires participation of either two living parents or at least one full sibling with diabetes. To be enrolled as having nephropathy, the diabetic sib must meet one of the following criteria:

* renal biopsy consistent with a diagnosis of diabetic nephropathy;
* urinary albumin excretion ≥ 30 mg/24hr or a urine albumin (mg/dl)/creatinine (mg/dl) ratio ≥ 0.03;
* a serum creatinine concentration ≥ 1.6 mg/dl for men or ≥ 1.4 mg/dl for women; or
* ESRD. Unaffected sibs are recruited if they have had diabetes for ≥ 10 years, have normal serum creatinine and albumin excretion (< 30 mg albumin/24 hours, or a urine albumin (mg/dl)/creatinine (mg/dl) ratio < 0.03) and no historical evidence of kidney disease.

The criteria for MALD control subjects differ by ethnic group. For the African-American MALD protocol, two different control samples are recruited. First, an adult offspring with or without renal disease and the other parent of the offspring, who cannot have evidence of renal disease, are collected as controls for African-American probands with either diabetic or non-diabetic nephropathy. Together with the probands, this forms a sample of triads (offspring and other parent) or dyads (spouse only). A second group of African-American control subjects consists of unrelated individuals with diabetes duration ≥ 10 years and without nephropathy (as defined above for diabetic sibs). For Mexican Americans, a single unrelated control population is recruited with diabetes duration ≥ 10 years but without nephropathy (as defined above for diabetic sibs).

Exclusion Criteria:

A. Did not sign the informed consent: refusal to participate. B. Diagnosis not confirmed. C. Appropriate siblings not available. D. Judged not likely or unable to follow study protocol. E. Ethnicity of parents or grandparent not suitable. F. Spouse not available.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9031 (Actual)
Dates: Start 1999-10 (Actual); Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sudha Iyengar, PhD, Principal Investigator — Case Western Reserve University; Barry I Freedman, MD, Study Chair — Wake Forest University; Sharon Adler, MD, Principal Investigator — University of California, Los Angeles; Hanna Abboud, MD, Principal Investigator — University of Texas Health Sciences Center at San Antonio; John R Sedor, MD, Principal Investigator — Case Western Reserve University; Rulan Parekh, MD, Principal Investigator — Johns Hopkins University; Philip Zager, MD, Principal Investigator — University of New Mexico; William Knowler, MD, PhD, Principal Investigator — NIDDK-Phoenix; Susanne Nicholas, MD, Principal Investigator — University of California, Los Angeles; Rebekah Rasooly, PhD, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK); Paul Kimmel, MD, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (5):
- United States (5):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California Los Angeles, Los Angeles, California
  - Harbor-UCLA Medical Center, Torrance, California
  - Johns Hopkins University, Baltimore, Maryland
  - Case Western Reserve University, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Data are available at the NIDDK Central Repository, https://repository.niddk.nih.gov/studies/find/
URL: https://repository.niddk.nih.gov/studies/find/

REFERENCES:
- [Background] Knowler WC, Coresh J, Elston RC, Freedman BI, Iyengar SK, Kimmel PL, Olson JM, Plaetke R, Sedor JR, Seldin MF; Family Investigation of Nephropathy and Diabetes Research Group. The Family Investigation of Nephropathy and Diabetes (FIND): design and methods. J Diabetes Complications. 2005 Jan-Feb;19(1):1-9. doi: 10.1016/j.jdiacomp.2003.12.007. PMID 15642484
- [Result] Bostrom MA, Kao WH, Li M, Abboud HE, Adler SG, Iyengar SK, Kimmel PL, Hanson RL, Nicholas SB, Rasooly RS, Sedor JR, Coresh J, Kohn OF, Leehey DJ, Thornley-Brown D, Bottinger EP, Lipkowitz MS, Meoni LA, Klag MJ, Lu L, Hicks PJ, Langefeld CD, Parekh RS, Bowden DW, Freedman BI; Family Investigation of Nephropathy and Diabetes (FIND) Research Group. Genetic association and gene-gene interaction analyses in African American dialysis patients with nondiabetic nephropathy. Am J Kidney Dis. 2012 Feb;59(2):210-21. doi: 10.1053/j.ajkd.2011.09.020. Epub 2011 Nov 25. PMID 22119407
- [Result] Iyengar SK, Abboud HE, Goddard KA, Saad MF, Adler SG, Arar NH, Bowden DW, Duggirala R, Elston RC, Hanson RL, Ipp E, Kao WH, Kimmel PL, Klag MJ, Knowler WC, Meoni LA, Nelson RG, Nicholas SB, Pahl MV, Parekh RS, Quade SR, Rich SS, Rotter JI, Scavini M, Schelling JR, Sedor JR, Sehgal AR, Shah VO, Smith MW, Taylor KD, Winkler CA, Zager PG, Freedman BI; Family Investigation of Nephropathy and Diabetes Research Group. Genome-wide scans for diabetic nephropathy and albuminuria in multiethnic populations: the family investigation of nephropathy and diabetes (FIND). Diabetes. 2007 Jun;56(6):1577-85. doi: 10.2337/db06-1154. Epub 2007 Mar 15. PMID 17363742
- [Result] Igo RP Jr, Iyengar SK, Nicholas SB, Goddard KA, Langefeld CD, Hanson RL, Duggirala R, Divers J, Abboud H, Adler SG, Arar NH, Horvath A, Elston RC, Bowden DW, Guo X, Ipp E, Kao WH, Kimmel PL, Knowler WC, Meoni LA, Molineros J, Nelson RG, Pahl MV, Parekh RS, Rasooly RS, Schelling JR, Shah VO, Smith MW, Winkler CA, Zager PG, Sedor JR, Freedman BI; Family Investigation of Nephropathy and Diabetes Research Group. Genomewide linkage scan for diabetic renal failure and albuminuria: the FIND study. Am J Nephrol. 2011;33(5):381-9. doi: 10.1159/000326763. Epub 2011 Mar 31. PMID 21454968
- [Result] Thameem F, Igo RP Jr, Freedman BI, Langefeld C, Hanson RL, Schelling JR, Elston RC, Duggirala R, Nicholas SB, Goddard KA, Divers J, Guo X, Ipp E, Kimmel PL, Meoni LA, Shah VO, Smith MW, Winkler CA, Zager PG, Knowler WC, Nelson RG, Pahl MV, Parekh RS, Kao WH, Rasooly RS, Adler SG, Abboud HE, Iyengar SK, Sedor JR; Family Investigation of Nephropathy and Diabetes Research Group. A genome-wide search for linkage of estimated glomerular filtration rate (eGFR) in the Family Investigation of Nephropathy and Diabetes (FIND). PLoS One. 2013 Dec 17;8(12):e81888. doi: 10.1371/journal.pone.0081888. eCollection 2013. PMID 24358131